CLINICAL TRIAL: NCT00599521
Title: A Multi-Center, Randomized, Double-Blind, Parallel Group Study to Demonstrate the Efficacy and Safety of Adapalene Lotion, 0.1% Compared With Vehicle Lotion in Subjects With Acne Vulgaris
Brief Title: Clinical Study to Test the Efficacy and Safety of Adapalene, 0.1%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Marie Ciardella Clinical Trials.gov Administrator, Galderma Laboratories, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.06.SPR.18114; IND 076057
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2011-03

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Adapalene
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adapalene lotion 0.1% (Experimental)
  Interventions: Drug: Adapalene lotion 0.1%
- Adapalene Lotion vehicle (Placebo Comparator)
  Interventions: Drug: Adapalene Lotion Vehicle

INTERVENTIONS:
Drug: Adapalene lotion 0.1% — Adapalene, 0.1% will be applied topically to the face, once a day, for 12 weeks
  Arms: Adapalene lotion 0.1%
Drug: Adapalene Lotion Vehicle — Vehicle will be applied topically to the face, once a day, for 12 weeks
  Arms: Adapalene Lotion vehicle

SUMMARY:
The purpose of this study is to determine whether Adapalene, 0.1% is safe and effective in the treatment of Acne Vulgaris.

DETAILED DESCRIPTION:
This study will compare the efficacy and safety of Adapalene, 0.1% and vehicle in the treatment of subjects with Acne Vulgaris. This is a multi-center, randomized, double-blind, parallel, vehicle controlled study involving subjects with acne vulgaris meeting pre-specified inclusion/exclusion criteria. Male and female subjects, 12 years of age or older, with 20-50 papules and pustules and 30 to 100 non-inflammatory lesions and have an Investigator's Global Assessment (IGA) score of 3 (Moderate) or 4 (Severe) are eligible for enrollment. One nodule may be present at inclusion. Acne lesions are evaluated on the face only. Subjects presenting with facial and truncal acne vulgaris can participate in this study. Subjects will be randomized in a 1:1 ratio to Adapalene, 0.1% or Vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Moderate or Severe Acne Vulgaris,
* 20-50 papules and pustules in total on the face excluding the nose
* 30-100 non-inflammatory lesions on the face excluding the nose.
* Negative urine pregnancy test for all females.

Exclusion Criteria:

* Subjects with more than one acne nodule.
* Subjects with any acne cyst on the face.
* Subjects with acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.), or severe acne requiring systemic treatment.
* Subjects with underlying diseases or other dermatologic conditions that require the use of interfering topical or systemic therapy, such as, but not limited to, atopic dermatitis, perioral dermatitis or rosacea.
* Subjects who are pregnant, nursing, or planning a pregnancy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1067 (Actual)
Dates: Start 2007-11; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (29):
  - University of California, San Diego, California
  - Dermatology Specialists, Inc., Vista, California
  - Cherry Creek Dermatology, Denver, Colorado
  - Advanced Dermatology and Cosmetic Surgery, Ormond Beach, Florida
  - Dermatology Research, Pinellas Park, Florida
  - Christie Clinic, PC, Champaign, Illinois
  - Compliant Clinical Research, Olathe, Kansas
  - Dermatology Specialists, Louisville, Kentucky
  - East Coast Clinical Research, Inc., Haverhill, Massachusetts
  - Midwest Cutaneous Research, Clinton Township, Michigan
  - Henry Ford Medical Center-Dept. of Dermatology, Detroit, Michigan
  - Minnesota Clinical Study Centert, Fridley, Minnesota
  - Skin Specialists, PC, Omaha, Nebraska
  - Cindy Lamerson, Reno, Nevada
  - Fran Cook-Bolden, New York, New York
  - Dermatology Associates of Rochester, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - University Dermatology Consultants, Cincinnati, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Northwest Cutaneous Research Specialists, Portland, Oregon
  - Palmetto Medical Research, Mt. Pleasant, South Carolina
  - Dermatology Associates, Knoxville, Tennessee
  - Dermatology Research Associates, Nashville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - J&S Studies, Inc., Bryan, Texas
  - The Center for Skin Research, Houston, Texas
  - Dermatology Research Center, Salt Lake City, Utah
  - Premier Clinical Research, Spokane, Washington
- Canada (5):
  - Dermatology Associates, Calgary, Alberta
  - Derm Research @ 888 Inc, Vancouver, British Columbia
  - Ultranova Skincare, Barrie, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Siena Medical Research, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multi center study recruitment period: First subject enrolled Nov 6, 2007; last subject completed Nov 14, 2008
Pre-assignment Details: Washout requirements: 2 weeks for systemic anti-inflammatory drugs, 4 weeks for oral antibiotics, 2 months for inhaled/nasal steroids and 6 months for hormonal contraceptives/therapies.
Groups:
- Adapalene Lotion 0.1%; Adapalene Lotion Vehicle 0%: once a day for 12 weeks
Period: Overall Study
Arm/Group | Adapalene Lotion 0.1% | Adapalene Lotion Vehicle 0%
Started | 535 | 531
Completed | 475 | 462
Not Completed | 60 | 69
Not completed — Lack of Efficacy | 4 | 8
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 28 | 34
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 23 | 23
Not completed — Pregnancy | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adapalene Lotion 0.1% | Adapalene Lotion Vehicle 0% | Total
Number analyzed (Participants) | 535 | 531 | 1066
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 338 | 336 | 674
  Between 18 and 65 years | 197 | 195 | 392
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.1 (6.8) | 19.2 (7.3) | 19.15 (7.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 300 | 272 | 572
  Male | 235 | 259 | 494
Region of Enrollment [Number; unit: participants]
  United States | 487 | 484 | 971
  Canada | 48 | 47 | 95

OUTCOME MEASURES:

1. Primary Outcome: Co-Primary Endpoint: Success Rate on Investigator's Global Assessment (IGA) From Baseline to Week 12
Description: Success defined as percentage of subjects who achieved at least a two-grade reduction in IGA scale (e.g from moderate to clear or almost clear)at week 12 from baseline, Last Observation Carried Forward, Intent to treat population. The IGA (Investigator Global Assessment) is defined as a 5 point scale (0 to 4). "0" = clear , "1"= almost clear, "2"= mild, "3"= moderate, "4"=severe.
Time Frame: From Baseline to Week 12
Measure: Number; unit: Percentage of Participants
Arm/Group | Adapalene Lotion 0.1% | Adapalene Lotion Vehicle 0%
Number analyzed (Participants) | 535 | 531
Percentage of Participants | 24.1 | 16.4

2. Primary Outcome: Co-Primary Endpoint: Absolute Change in Total Lesion Counts From Baseline to Week 12
Time Frame: Baseline to 12 weeks
Measure: Least Squares Mean (Standard Error); unit: Absolute Change in Total Lesion Count
Arm/Group | Adapalene Lotion 0.1% | Adapalene Lotion Vehicle 0%
Number analyzed (Participants) | 535 | 531
Absolute Change in Total Lesion Count | 32.5 (1.0) | 23.3 (1.0)

3. Secondary Outcome: Mean Percent Change in Total Lesion Count From Baseline to Week 12
Description: Percent change in lesion count from baseline to week 12
Time Frame: From Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: % Change in Lesion Count
Arm/Group | Adapalene Lotion 0.1% | Adapalene Lotion Vehicle 0%
Number analyzed (Participants) | 535 | 531
% Change in Lesion Count
  Total lesion count | -44.6 (33.2) | -32.8 (34.1)
  Inflammatory | -46.0 (36.8) | -36.9 (40.7)
  Non-Inflammatory | -43.1 (40.9) | -30.2 (40.5)

4. Primary Outcome: Co-Primary Endpoint: Absolute Change in Inflammatory Lesion Count From Baseline to Week 12
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Absolute Change in Infl Lesion count
Arm/Group | Adapalene Lotion 0.1% | Adapalene Lotion Vehicle 0%
Number analyzed (Participants) | 535 | 531
Absolute Change in Infl Lesion count | 13.0 (0.5) | 10.4 (0.5)

5. Primary Outcome: Co-Primary Endpoint: Absolute Change in NonInflammatory Lesion Counts From Baseline to Week 12
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Absolute Change in Non-Infl Lesion
Arm/Group | Adapalene Lotion 0.1% | Adapalene Lotion Vehicle 0%
Number analyzed (Participants) | 535 | 531
Absolute Change in Non-Infl Lesion | 19.5 (0.8) | 12.9 (0.8)

ADVERSE EVENTS:
Arm/Group | Adapalene Lotion 0.1% | Adapalene Lotion Vehicle 0%
Serious Adverse Events (participants affected / at risk) | 0/535 | 0/531
Other Adverse Events (participants affected / at risk) | 32/535 | 11/531
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene Lotion 0.1% (N=535) | Adapalene Lotion Vehicle 0% (N=531)
Dry Skin (Skin and subcutaneous tissue disorders) | 32 (33) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
disclosure restriction varies per institutional request/agreement